CLINICAL TRIAL: NCT06709963
Title: The Effect of Intermittent Theta Burst Stimulation on Brain Characteristics, Pain Intensity, and Cognitive Functions in Older People with Chronic Musculoskeletal Pain: a Double-blinded, Randomized, Sham-controlled, Mixed-methods, Pilot Trial with a Six-month Post-treatment Follow-up.
Brief Title: The Effect of Intermittent Theta Burst Stimulation on Brain Characteristics, Pain Intensity, and Cognitive Functions in Older People with Chronic Musculoskeletal Pain.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Arnold Wong Yu Lok, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20240411013
Record Dates: First submitted 2024-11-22; First posted 2024-11-29 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Chronic Non-Specific Low Back Pain; Chronic Knee Pain; Chronic Musculoskeletal Pain
Keywords: Chronic non-specific low back pain; rTMS; Sham; Chronic knee pain; DLPFC; chronic musculoskeletal pain; iTBS

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Sham (Sham Comparator)
  Interventions: Device: ITBS
- Left DLPFC (Experimental)
  Interventions: Device: ITBS

INTERVENTIONS:
Device: ITBS — We will use a coil called Cool-6000 A/P to conduct real and sham control. This coil will be placed on the scalp of older adults. The iTBS protocol will begin with a 2-s burst train (totally 30 pulses), repeating every 10 s. Each burst train will consist of 10 triplet pulses with an inter-burst interval of 0.16 s, thus the triplets fire at a rate of 5 Hz. ITBS parameters will include three continuous pulses at 50 Hz repeated at 5 Hz (2s on, 8s off) for a total of 600 pulses.
  We will administer two rounds of iTBS per treatment day, with a 15-minute interval between the two sessions. In total, each participant will receive 1,200 stimuli during a single-session iTBS, totaling for 14 days. Each treatment session will last for about 30 minutes. Intermittent θ-burst stimulation intensity will be set at 70% of the resting motor threshold.

SUMMARY:
The goal of this clinical trial is to explore the effects of accelerated intermittent Theta Burst Stimulation (iTBS) on pain relief and cognitive function in older adults with chronic musculoskeletal pain. It will also utilize magnetic resonance imaging to illustrate the neurophysiological mechanisms underlying the role of iTBS in improving various outcome indicators in this population.

The main questions it aims to answer are:

1. Is left dorsolateral prefrontal cortex stimulation using accelerated iTBS effective for older adults with chronic musculoskeletal pain?
2. What are the neurophysiological mechanisms underlying the role of iTBS in improving various outcome indicators in older adults with chronic musculoskeletal pain?

Participants will:

1. Receive 1,200 stimuli during a single-session iTBS, totaling 14 days.
2. Undergo MRI scanning before, immediately after treatment, cognitive and pain-related tests before, immediately after treatment, and during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* have normal cognitive function (Hong Kong Montreal Cognitive Assessment ≥ 26)
* be right-handed
* be able to speak Cantonese
* chronic nonspecific low back pain, or having both chronic nonspecific low back pain and chronic knee pain that has lasted for at least 3 months
* an average pain intensity of ≥ 5 out of 10 on an 11-point numerical rating scale in the last 7 days, where 0 means "no pain" and 10 means "worst pain imaginable"
* having pain at least half of the days in the past 4 weeks.
* have at least 6 years of formal education and know how to read and write Chinese
* agree to sign an informed consent and complete the experiment tests
* be able to communicate via email or text message, as several study measures will be collected electronically

Exclusion Criteria:

* inability to ambulate without assistance from another person (canes or walkers will be allowed);
* having specific causes of chronic nonspecific low back pain, or having both chronic nonspecific low back pain and chronic knee pain (e.g., spinal stenosis, lumbar disc herniation, spondylolisthesis, recent vertebral fracture, spinal infection);
* having other concurrent musculoskeletal conditions at other body parts (e.g., fibromyalgia, or neck pain)
* self-reported history of lumbar or lower extremity surgery
* self-reported history of neurological or psychiatric disorders (e.g., stroke, brain surgery, head trauma; schizophrenia, multiple personality disorder, dissociative identity disorder, stroke) or self-reported cancer history
* self-reported specific inflammatory disorder: rheumatoid arthritis, rheumatica, scleroderma, lupus, or polymyositis
* unexplained, unintended weight loss of 20 lbs or more in the past year
* cauda equina syndrome
* uncorrected visual deficit
* drug or alcohol addiction
* taken alcohol, opioids or benzodiazepines medicines 24 hours before the experiment
* claustrophobia
* contraindications for undergoing the magnetic resonance imaging (MRI) examination based on the MRI safety screening form of University Research Facility in Behavioral and Systems Neuroscience (UBSN) at The Hong Kong Polytechnic University (PolyU)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The recruitment rate, retention rate (completion rate), non-completion reasons, drop-out rate | Immediately after the intervention
  The recruitment rate, retention rate (completion rate), non-completion reasons, drop-out rate will be evaluated as our primary outcomes, because of the feasibility of the study.
ITBS acceptability questionnaire | Immediately after the intervention
  ITBS acceptability questionnaire has ten items of positive acceptability, ranged from 10 to 50, and it also has five items of negative acceptability, ranged from 5 to 25. The iTBS acceptability questionnaire has a total score ranging from 15 to 75.
Pain intensity assessment | Baseline, immediately after the intervention, five-month follow-up at one-month,three-month,six-month follow-up timepoints.
  The 11-point numerical rating scale, ranged from 0 to 10, higher scores indicate higher pain intensity.

SECONDARY OUTCOMES:
Depression, anxiety, and stress test | Baseline
  The Chinese version of the short Depression Anxiety Stress Scales, scores ranged from 0 to 13, higher scores for each domain (depression, anxiety, and stress) indicate more respective problems.
Disability evaluation | Baseline, immediately after the intervention, five-month follow-up at one-month,three-month,six-month follow-up timepoints.
  The Hong Kong Chinese Version of the Roland-Morris Disability Questionnaire has 24 items. Scores ranged from 0 to 24, higher scores indicate worse disability.
Pain catastrophizing assessment | Baseline, immediately after the intervention, five-month follow-up at one-month,three-month,six-month follow-up timepoints.
  The Chinese version of Pain Catastrophizing Score. The scores ranged from 0 to 13, higher scores indicate more pain catatrophizing thought.
Pain drawing test | Baseline
  The body map scoring system indicates the location of participants' painful site
Frailty status assessment | Baseline, immediately after the intervention, one-month follow-up timepoint.
  Fatigue, Resistance, Ambulation, Illness, and Loss, the presence of 3 of 5 item characteristics indicate the presence of frailty, scores ranged from 0 to 5. Lower scores mean more frailty.
Physical activity assessment | Baseline, immediately after the intervention, one-month follow-up timepoint.
  Physical Activity Scale for the Elderly; it has 3 domains (leisure, household, and occupation activities) to measure physical activity levels of adults aged 65 or above. higher scores indicate more active.
Sleep quality assessment | Baseline, immediately after the intervention, one-month follow-up timepoint.
  Pittsburgh Sleep Quality Index. It has 7 domains to measure sleep quality , sleep latency, sleep duration, habital sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Scores ranged from 0 to 21, higher scores indicate poorer sleep quality.
Cognitive function screening | Baseline
  Hong Kong Montreal Cognitive Assessment. It is a cognitive screening tool specifically adapted for Chinese older adults in Hong Kong. It is designed to detect mild cognitive impairment and dementia. A score < 26 suggests participant has mild cognitive impairment.
Working memory test inside magnetic resonance imaging scanning | Baseline, immediately after the intervention
  The digit 2-back task, more response accuracy of digits indicates better working memory
Cognitive flexibility test inside magnetic resonance imaging scanning | Baseline, immediately after the intervention.
  The More Odd Shifting task, It requires participants to switch between different mental sets or rules, such as identifying odd numbers or shifting between different categories. Better response accuracy indicates better cognitive flexibility
Cognitive inhibition test inside magnetic resonance imaging scanning | Baseline, immediately after the intervention.
  Color-Word Matching Stroop Task, more correct matching indicate better ability to inhibit cognitive interference
Perseveration and abstract reasoning test outside magnetic resonance imaging scanning | Baseline, immediately after the intervention, one-month follow-up timepoint.
  The Modified Wisconsin Card Sorting Test, more correct matching of cards indicate better perseveration and abstract reasoning.
Working memory Test outside magnetic resonance imaging scanning | Baseline, immediately after the intervention, one-month follow-up timepoint.
  The Verbal Digits Forward and Backward Test, more correct recall of digits indicate better working memory and executive function
Cognitive flexibility test outside magnetic resonance imaging scanning | Baseline, immediately after the intervention, one-month follow-up timepoint.
  The Trail Making Tests, a neuropsychological test of visual attention and task switching, completing the trail correctly within a shorter period of time means better cognitive flexibility
Inhibition test outside magnetic resonance imaging scanning | Baseline, immediately after the intervention, one-month follow-up timepoint.
  Go/NoGo task, more response accuracy indicates better control of inhibition.

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Dr WONG, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No